CLINICAL TRIAL: NCT02792309
Title: Strengthening Relationship Education and Marriage Services - Impact Evaluation of MotherWise Program
Brief Title: Impact Evaluation of MotherWise Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MPR-50098-UD
Record Dates: First submitted 2016-05-25; First posted 2016-06-07 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-02

CONDITIONS: Parenting; Family Relations; Marriage; Mother-Child Relations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MotherWise Programming (Experimental): Three components: (1) 18 hours of core workshop sessions using the Within My Reach relationship education curriculum supplemented with content on mother-infant relationships; (2) case management services; and (3) optional relationship education workshops for couples.
  Interventions: Behavioral: MotherWise Program
- Control (No Intervention): No program services

INTERVENTIONS:
Behavioral: MotherWise Program — Healthy Marriage or Relationship Education services for pregnant women.
  Arms: MotherWise Programming

SUMMARY:
Mathematica was awarded a contract by ACF to conduct the evaluation of selected grantees offering Healthy Marriage and Relationship Education Programs.This particular evaluation will focus on the University of Denver's MotherWise program, which offers relationship education and other supports to low-income women expecting a baby. The program has three core components: (1) 18 hours of core workshop sessions using the Within My Reach relationship education curriculum supplemented with content on mother-infant relationships; (2) case management services; and (3) optional relationship education workshops for couples. The evaluation will test the effect of this full package of services on mothers' relationship outcomes, as well as other outcomes related to child well-being, such as co-parenting and father involvement.

DETAILED DESCRIPTION:
The U.S. Department of Health and Human Services (HHS), Administration for Children and Families (ACF), is conducting an evaluation of healthy marriage and relationship education (HMRE) programs. Mathematica was awarded a contract by ACF to conduct the evaluation of selected programs/grantees.This segment of the larger evaluation will focus on the University of Denver's MotherWise program.

The Mother Wise program will offer relationship education and other supports to low-income women expecting a baby. The program will have three core components: (1) 18 hours of core workshop sessions using the Within My Reach relationship education curriculum supplemented with content on mother-infant relationships; (2) case management services; and (3) optional relationship education workshops for couples. The evaluation will test the effect of this full package of services on mothers' relationship outcomes, as well as other outcomes related to child well-being, such as co-parenting and father involvement. If feasible, the evaluation will also examine some measures available through hospital records, such as birth weight.

Mother Wise will enroll women who are expecting a baby and those who have had a baby within the past month.

Control group members will not be eligible for Mother Wise but will be eligible for other services available in the community.

To document the outcomes of study participants, survey data will be collected at two time points: (1) a baseline survey administered at study enrollment, a (2) a 12-month follow-up survey, and (3) a 30-month follow-up survey. Surveys will be conducted by staff at Mathematica's Survey Operations Center using computer-assisted telephone interviewing (CATI). Survey data may be supplemented with administrative records data from the Denver Health system.

ELIGIBILITY:
Inclusion Criteria:

To be eligible, women must be expecting a baby or had a baby in the past 3 months.

Exclusion Criteria:

To be eligible, women must not be incarcerated.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 953 (Actual)
Dates: Start 2016-09; Primary Completion 2021-09 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Perceived romantic relationship skills | 1 year after random assignment
  Six-item scale (ranges from 1 to 4)
Perceived romantic relationship skills | 30 months after random assignment
  Six-item scale (ranges from 1 to 4)
Perceived conflict management skills | 1 year after random assignment
  Five-item scale (ranges from 1 to 4)
Perceived conflict management skills | 30 months after random assignment
  Five-item scale (ranges from 1 to 4)
Support for going slow in romantic relationships | 1 year after random assignment
  One-item scale (ranges from 1 to 4)
Support for going slow in romantic relationships | 30 months after random assignment
  One-item scale (ranges from 1 to 4)
Disapproval of couple violence | 1 year after random assignment
  Five-item scale (ranges from 1 to 4)
Disapproval of couple violence | 30 months after random assignment
  Five-item scale (ranges from 1 to 4)
Any psychological abuse | 1 year after random assignment
  A binary variable equal to 1 if the mother indicates that a romantic partner has subjected her to psychological abuse in the past year.
Any psychological abuse | 30 months after random assignment
  A binary variable equal to 1 if the mother indicates that a romantic partner has subjected her to psychological abuse in the past year.
Any physical abuse | 1 year after random assignment
  A binary variable equal to 1 if the mother indicates that a romantic partner has pushed, shoved, kicked, punched or beaten her up in the past year.
Any physical abuse | 30 months after random assignment
  A binary variable equal to 1 if the mother indicates that a romantic partner has pushed, shoved, kicked, punched or beaten her up in the past year.
Had an unintended pregnancy since program enrollment | 1 year after random assignment
  A binary variable equal to 1 if the mother reported having had an unintended pregnancy since random assignment.
Had an unintended pregnancy since program enrollment | 30 months after random assignment
  A binary variable equal to 1 if the mother reported having had an unintended pregnancy since random assignment.
Quality of co-parenting relationship with baby's father | 1 year after random assignment
  Ten-item scale (ranges from 0 to 10)
Quality of co-parenting relationship with baby's father | 30 months after random assignment
  Ten-item scale (ranges from 0 to 10)
Depressive symptoms | 1 year after random assignment
  Eight-item scale (ranges from 0 to 24; based on PHQ-8)
Depressive symptoms | 30 months after random assignment
  Eight-item scale (ranges from 0 to 24; based on PHQ-8)
Number of relationship transitions | 30 months after random assignment
  This is a continuous variable representing the number of relationship transitions the mother reported since random assignment. A relationship transition occurs each time a romantic relationship begins or ends.
Material hardship | 30 months after random assignment
  This continuous variable ranges from 0 to 6 and reflects how many of six possible things a mother had done in the past year because she did not have enough money.
Child social-emotional and behavioral problems | 30 months after random assignment
  This 31-item scale is a measure of the child's social-emotional and behavioral problems with higher scores indicating more problems.
Child social-emotional abilities | 30 months after random assignment
  This 11-item scale is a measure of the child's social-emotional abilities-such as empathy, prosocial behaviors, and compliance-with higher scores indicating higher competence.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wood, PhD, Principal Investigator — Mathematica Policy Research
Locations (1):
- University of Denver, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Restricted use files will be made available to researchers via the Inter-University Consortium for Political and Social Research (ICPSR) at the University of Michigan
Time Frame: Mid-2022
Access Criteria: Yet to be determined

REFERENCES:
- [Derived] Mazzoni SE, O'Reilly Treter M, Hyer J, Pena R, Rhoades GK. Impact of Prenatal Group Healthy Relationship Education on Postpartum Contraception. Womens Health Rep (New Rochelle). 2023 Mar 27;4(1):148-153. doi: 10.1089/whr.2022.0104. eCollection 2023. PMID 37008185